CLINICAL TRIAL: NCT01557283
Title: An Observational Study of the Real Life Management of the Psoriasis Patients Treated With Enbrel According to the New Reimbursement Criteria - Beflex Study
Brief Title: An Observational Study of the Real Life Management of the Psoriasis Patients Treated With Enbrel According to the New Reimbursement Criteria
Acronym: BEFLEX
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801314; BEFLEX
Record Dates: First submitted 2011-09-30; First posted 2012-03-19 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-05

CONDITIONS: Plaque Psoriasis Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Plaque psoriasis patients: Plaque psoriasis patients treated with Enbrel after the approval of the new belgian reimbursement criteria
  Interventions: Other: Enbrel treatment

INTERVENTIONS:
Other: Enbrel treatment — Enbrel SC 50mg once weekly or 25mg twice weekly

SUMMARY:
With the new reimbursement criteria, we want:

To describe the average treatment duration of patients with Enbrel expressed as a number of weeks/year.

To describe the number of patients who receive continuous treatment To describe the number of patients who receive intermittent treatment To describe the number of weeks off treatment

DETAILED DESCRIPTION:
100 patients will be followed for at least 1 year

ELIGIBILITY:
Inclusion Criteria:

* Patient restarts or is starting treatment with Enbrel for his/her psoriasis in alignment with reimbursement criteria
* Patients ≥18 year
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects enrolled should meet the usual prescribing criteria for Enbrel as per local reimbursement criteria and should be entered into the study at the investigator's discretion. It is requested to include patients in a consecutive manner as much as possible.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Herestraat 49, Leuven, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801314&StudyName=An%20Observational%20Study%20of%20the%20Real%20Life%20Management%20of%20the%20Psoriasis%20Patients%20Treated%20with%20Enbrel%20According%20to%20the%20New%20Reimbursement%20Cr

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants who had moderate to severe plaque psoriasis and received etanercept (Enbrel) as per Summary of Product Characteristics (SmPC), were observed for at least 1 year. According to SmPC, recommended dose included etanercept 25 milligram (mg) twice weekly or 50 mg once weekly subcutaneous injection. Participants either received etanercept in treatment cycles of up to 24 weeks with at least 2 weeks of treatment discontinuation between the cycles or continuously without any treatment discontinuation as per dermatologist's discretion.
Period: Overall Study
Arm/Group | Etanercept
Started | 140
Completed | 96
Not Completed | 44
Not completed — Lost to Follow-up | 7
Not completed — Non-responder | 19
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 1
Not completed — Non-compliance | 1
Not completed — Withdrawal by Subject | 1
Not completed — Participant's weight too high for dose | 1
Not completed — Worsening of psoriasis | 1
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Per protocol (PP) population included participants who completed at least 1 treatment cycle, for whom study conclusion was duly filled in, and who had not deviated from protocol.
Arm/Group | Etanercept
Number analyzed (Participants) | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.83 (12.428)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Weeks of Etanercept Treatment
Description: Average duration of time in weeks for treatment with etanercept was reported.
Time Frame: Baseline up to end of study (90 weeks)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 138
weeks | 48.1874 (17.55204)

2. Secondary Outcome: Number of Weeks of Off-Treatment
Description: Total duration of time in weeks for which participants discontinued etanercept treatment was reported.
Time Frame: Baseline up to end of study (90 weeks)
Population: Per protocol (PP) population included participants who completed at least 1 treatment cycle, for whom study conclusion was duly filled in, and who had not deviated from protocol. Here 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 121
weeks | 5.5348 (10.15699)

3. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score
Description: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 sections: head, arms, trunk, and legs. For each section, percent (%) area of skin involved was estimated: 0 = 0%, 1 = less than (<) 10%, 2 = 10 to <30%, 3 = 30 to <50%, 4 = 50 to <70%, 5= 70 to <90%, 6 = 90 to 100%. Severity was estimated by clinical signs: erythema, induration, desquamation; scale: 0 = none to 4 = maximum. Final PASI = sum of severity parameters for each section*area score*weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4); total possible score range: 0= no disease to 72= maximal disease.
Time Frame: Start and end of cycle 1, 2, 3
Population: Per protocol (PP) population included participants who completed at least 1 treatment cycle, for whom study conclusion was duly filled in, and who had not deviated from protocol. 'N' (number of participants analyzed) signifies participants evaluable for this measure; 'n' signifies participants evaluable for this measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 136
units on a scale
  Start of Cycle 1 (n=136) | 10.913 (8.6412)
  End of Cycle 1 (n=123) | 6.680 (7.6061)
  Start of Cycle 2 (n=114) | 6.395 (6.1129)
  End of Cycle 2 (n=87) | 5.571 (6.0198)
  Start of Cycle 3 (n=81) | 5.504 (5.3579)
  End of Cycle 3 (n=25) | 5.468 (6.2810)

4. Secondary Outcome: Percentage of Body Surface Area (BSA) Affected by Psoriasis
Description: Percentage of body surface area affected by psoriasis was estimated using the palm method: one of the participant's palm to proximal interphalangeal and thumb = 1 percent (%) of total BSA. Regions of the body were assigned specific number of palms with percentage [Head and neck = 10% (10 palms), upper extremities = 20% (20 palms), Trunk (axillae and groin) = 30% (30 palms), lower extremities (buttocks) = 40% (40 palms)]. The total BSA affected was the summation of individual regions affected.
Time Frame: Start and end of cycle 1, 2, 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Etanercept
Number analyzed (Participants) | 129
percentage of BSA
  Start of Cycle 1 (n=129) | 14.189 (14.8781)
  End of Cycle 1 (n=115) | 8.016 (10.8758)
  Start of Cycle 2 (n=108) | 7.579 (8.8944)
  End of Cycle 2 (n=84) | 5.361 (5.9864)
  Start of Cycle 3 (n=78) | 5.706 (6.9649)
  End of Cycle 3 (n=28) | 10.221 (16.3993)

5. Secondary Outcome: Number of Participants With Reasons for Treatmant Discontinuation
Description: Number of participants who discontinued etanercept before completing the study was reported.
Time Frame: Baseline up to end of study (90 weeks)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 138
participants
  Non-responders | 19
  Adverse Event | 7
  Lack of Efficacy | 1
  Non-compliance | 1
  Withdrawal by Subject | 1
  Participant's weight too high for dose | 1
  Worsening of Psoriasis | 1
  Unspecified | 1

6. Other Pre Specified Outcome: Number of Participants Who Received Continuous Treatment
Description: Number of participants who were treated continuously with etanercept without any treatment discontinuation as per dermatologist's discretion was reported.
Time Frame: Baseline up to end of study (90 weeks)
Population: Per protocol (PP) population included participants who completed at least 1 treatment cycle, for whom study conclusion was duly filled in, and who had not deviated from protocol. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 121
participants | 80

7. Other Pre Specified Outcome: Number of Participants Who Received Intermittent Treatment
Description: Number of participants who received etanercept treatment in cycles of up to 24 weeks with at least 2 weeks of treatment discontinuation was reported.
Time Frame: Baseline up to end of study (90 weeks)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 121
participants | 41

ADVERSE EVENTS:
Description: Same event may appear as both AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 subject and as nonserious in another subject, or 1 subject may have experienced both serious and nonserious event during study. All participants included in per protocol population were evaluable for safety.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 7/138
Other Adverse Events (participants affected / at risk) | 28/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=138)
Cholecystolithiasis (Hepatobiliary disorders) | 1
Obesity and surgery (Metabolism and nutrition disorders) | 1
Paget's disease (Musculoskeletal and connective tissue disorders) | 1
Breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Respiratory tract infection viral (Respiratory, thoracic and mediastinal disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Intervertebral disc operation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=138)
Lymphocytosis (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Functional digestive disorders, not elsewhere classified (Gastrointestinal disorders) | 1
Injection site reaction (General disorders) | 2
Leg edema (General disorders) | 1
Face edema (General disorders) | 1
Fatigue (General disorders) | 1
Hepatic dysfunction NOS (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Sinusitis (Infections and infestations) | 2
Rhinopharyngitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Weight loss (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Cluster headache (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Influenza (Respiratory, thoracic and mediastinal disorders) | 6
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Keratoacanthoma (Skin and subcutaneous tissue disorders) | 1
Ankle ulcer (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Furuncle (Skin and subcutaneous tissue disorders) | 1
Plastic operation on nose (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 1
Blood pressure high (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.